CLINICAL TRIAL: NCT05987293
Title: Mechanism and Risk Factors of Tracheal Tube-related Tongue Injury
Brief Title: A Single-center, Prospective Study for Mechanism and Risk Factors of Tracheal Tube-related Tongue Injury
Status: Active, not recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Li Fang Wang, attending doctor, China-Japan Friendship Hospital
Other Study IDs: ChinaJapanFHAnesth
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Tracheal Tube-related Tongue Injury
Keywords: intubation; general anesthesia; endotracheal intubation; post extubation dysphagia; post extubation stridor; tongue edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Supine group: Fifty-four patients undergoing elective surgery in general anesthesia for more than 2 hours with endotracheal tube applied in China-Japan Friendship Hospital will be enrolled (See in Sample Size calculation). Patients will be divided into two groups according to the surgery: supine position (Supine group)
  Interventions: Device: Tracheal tube-tongue pressure is measured using a computerized occlusal analysis system based on T-Scan® technique, suitable for multi-point real-time monitoring of intraoral pressure.
- Flexion group: The high-risk positions (Flexion group) which include patients scheduled for surgery under the prone position, cervical traction position, and beach chair position.
  Interventions: Device: Tracheal tube-tongue pressure is measured using a computerized occlusal analysis system based on T-Scan® technique, suitable for multi-point real-time monitoring of intraoral pressure.

INTERVENTIONS:
Device: Tracheal tube-tongue pressure is measured using a computerized occlusal analysis system based on T-Scan® technique, suitable for multi-point real-time monitoring of intraoral pressure. — A flexible film sensor with a thickness of 0.11mm is placed between the tongue and the tracheal tube to measure the distribution, join force and dynamic changes of pressure at different site of the tongue. Five channels of pressure values will be recorded separately: (Ch1) the tip of the tongue, (Ch2) the middle of the tongue, (Ch3) the base of the tongue, (Ch4) the right side at the base of the tongue, (Ch5) the left side at the base of the tongue. The pressure values at the following points during the operation will be recorded: (t1) after intubation, (t2) highest pressure during patient positioning, (t3) after position fixed, (t4) at the end of surgery, (t5) before extubation.

SUMMARY:
Article Summary

1. Tracheal tube-related tongue injury is a common clinical complication that would lead to serious events such as dysphagia, respiratory dysfuncion and macroglossia.
2. There is a lack of qualitative and quantitative risk assessment of tracheal tube-related tongue injury.
3. This is a protocol of a single-center, prospective, paralled-group clinical trial based on the measurement of dynamic changes in pressure between the tracheal tube and the tongue in different position during the surgery.
4. The primary endpoint is tracheal tube-related tongue injury, secondary outcomes include the time to first successful recovery of oral intake of fluids and solid food and airway-related events.
5. This trial aims to find the best indicators for tracheal tracheal tube-related tongue injury and to provide solid basis for optimizing airway protection strategies and surgical positioning.

DETAILED DESCRIPTION:
Background Tracheal tube-related tongue injury can lead to post-intubation pharyngeal dysfunction, postoperative macroglossia, or stridor after extubation. Possible mechanisms include increased oral pressure, obstruction of venous and lymphatic return in the neck, leading to severe throat pain, dysphagia, and respiratory function impairment. There is a lack of indicators and clinical awareness of this issue. Therefore we have designed this study to accurately monitor the tracheal tube-tongue pressure in different surgical position during general anesthesia.

Method This is a prospective, single-center observational study. Fifty-four patients undergoing elective surgery in general anesthesia for more than 2 hours with endotracheal tube applied will be enrolled. Patients will be divided into supine position (Supine group) and the high-risk positions (Flexion group) groups. Dynamic changes in pressure between the tracheal tube and the tongue are measured. All patients will be followed up until 7 days after operation. Primary endpoint is tracheal tube-related tongue injury. Secondary outcomes include the time to first successful recovery of oral intake of fluids and solid food, and airway-related events.

Discussion The study aims to explore the risk factors and pressure thresholds for tracheal tracheal tube-related tongue injury.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I-III
2. Age 18-85 years old
3. Scheduled for elective surgery with tracheal intubation under general anesthesia, with operation duration ≥2 hours
4. The intended surgical position will be supine, prone, cervical traction or beach chair position
5. Obtained informed consent

Exclusion Criteria:

1. Informed consent is not obtained
2. Maxillofacial surgeries or other surgeries involving the oral cavity and upper airway
3. History of head and neck radiotherapy
4. Deformity, trauma, infection and active bleeding exist in the mouth and tongue
5. Airway hyperresponsiveness, active asthma, acute exacerbation of chronic obstructive pulmonary disease, laryngeal osteomalacia
6. Respiratory insufficiency, moderate to severe ventilation or diffusion dysfunction
7. Existing chronic sore throat, recurrent laryngeal nerve injury, dysarthria, dysphagia, severe gastroesophageal reflux, upper esophageal sphincter dysfunction, cardiac stenosis and other basic diseases
8. Postoperative total parenteral nutrition therapy is planned

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty-four patients undergoing elective surgery in general anesthesia for more than 2 hours with endotracheal tube applied in China-Japan Friendship Hospital will be enrolled (See in Sample Size calculation). Patients will be divided into two groups according to the surgery: supine position (Supine group) and the high-risk positions (Flexion group) which include the prone position, cervical traction position, and beach chair position. Patients with existing oral or airway problems, or other factors influence postoperative recovery of diet will be excluded.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
tracheal tube-related tongue injury | Starting from the time after surgery till post-operative day 7 (POD7)
  The primary composite endpoint is assessed as incidence of tracheal tube-related tongue injury, which is either the state of severe sore throat (VAS≥4), dysphagia after extubation, or any of the symptoms of macroglossia.

SECONDARY OUTCOMES:
time of first smooth water intake | Starting from the time after surgery till post-operative day 7 (POD7)
  time of first smooth water intake
time of first smooth solid food intake | Starting from the time after surgery till post-operative day 7 (POD7)
  time of first smooth solid food intake
airway related events | Starting from the time after surgery till post-operative day 7 (POD7)
  bronchospasm, aspiration, secondary intubation, respiratory tract infection, respiratory insufficiency, prolonged oxygen therapy, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia Li, MD, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The original data of this trial include Case Record Form (CRF) and electronic data capture (EDC). Informed consent forms with patients' signature will be stored in private database for clinical trial in the department of anesthesiology. Electronic information will be stored in authorized computer following clinical trial confidentiality. Patient records are available from GOODWILL Electronic Medical Record System (Version 6.0) with medical access only. Test data related to this trial will be uploaded to http://www.medresman.org.cn/ within 2 weeks after collection, available to be public.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The original data of this trial include Case Record Form (CRF) and electronic data capture (EDC). Informed consent forms with patients' signature will be stored in private database for clinical trial in the department of anesthesiology. Electronic information will be stored in authorized computer following clinical trial confidentiality. Patient records are available from GOODWILL Electronic Medical Record System (Version 6.0) with medical access only. Test data related to this trial will be uploaded to http://www.medresman.org.cn/ within 2 weeks after collection, available to be public.
Access Criteria: http://www.medresman.org.cn/

REFERENCES:
- [Derived] Wang LF, Zheng MT, Liang N, Ma HN, Li WX. Study of postoperative laryngopharyngeal discomfort: protocol for a single-centre cohort study. BMJ Open. 2024 Jan 2;14(1):e079841. doi: 10.1136/bmjopen-2023-079841. PMID 38167285